CLINICAL TRIAL: NCT01291511
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate Prevention of Relapse in Patients With Schizophrenia Receiving Either Flexible Dose Iloperidone or Placebo in Long-term Use (up to 26 Weeks) Followed by up to 52 Weeks of Open-label Extension
Brief Title: Relapse Prevention Study in Patients With Schizophrenia
Acronym: REPRIEVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CILO522D2301
Record Dates: First submitted 2011-02-03; First posted 2011-02-08 (Estimated); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Mental Disorders; Antipsychotic Agents; Iloperidone; Relapse Prevention
MeSH Terms: conditions — Schizophrenia; Mental Disorders | interventions — iloperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Iloperidone (Experimental): After meeting all entry criteria, completing a 1-week open-label iloperidone titation period (up to 12 mg/day), followed by a 14-24 week open-label iloperidone flexible dose-stabilization period (up to 24 mg/day), approximately 260 patients will be randomized to one of two arms in a 1:1 ratio of iloperidone (flexible dosing 8-24 mg/day) to placebo. Post-randomization double-blind study medication will be administered orally twice daily for up to 26 weeks to evaluate relapse prevention. Subsequently, during the extension period, after a 1-week mock double-blind titration, open-label iloperidone (8-24 mg/day) is administered for up to 51 weeks to evaluate long-term safety.
  Interventions: Drug: Iloperidone
- Placebo (Placebo Comparator): Post-randomization matching placebo is administered orally bid during the double-blind period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iloperidone — Over-encapsulated iloperidone tablets were administered orally using a bid schedule; the strengths used include 1, 2, 4, 6, 8, 10, and 12 mg.
  Other Names: Fanapt®
  Arms: Iloperidone
Drug: Placebo — Matching placebo capsules were administered orally using a bid schedule during the double-blind period.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Iloperidone is effective in the prevention of relapse in patients with schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Patients must understand and be capable to communicate adequately with the study coordinator and to participate in cognitive testing.
* Patients must agree to cooperate with all tests and examinations required by the protocol, be willing to comply fully with treatment and able to ingest oral medication.
* Patients must understand the nature of the study and must sign an informed consent document.
* Patients will have a clear diagnosis of schizophrenia according to DSM-IV criteria for at least 1 year.
* Patients must need of ongoing psychiatric treatment and must have a documented reason why a change in treatment is needed which might lead to a clinical improvement
* At screening patients will have a Positive and Negative Syndrome Scale (PANSS) of no more than 100 and a Clinical Global Impression Scale (CGI) of no more than 5 (i.e. must not be severely ill or worse).
* Patients must be outpatients at the time of screening and have not been an inpatient to treat schizophrenia for at least 1 week prior to the screening visit.
* Patients must have a history of at least 2 prior episodes of relapse or impending relapse in the 2 years preceding the screening visit.

Exclusion Criteria:-

* Pregnant or nursing (lactating) women, or women who plan on conceiving during the course of the study.
* Patients who meet the DSM-IV criteria for schizophreniform disorder (295.40) and schizoaffective (295.70).
* Patients with active symptoms of any other primary psychiatric diagnosis (Axis I) or prominent Axis II disorder which would interfere with compliance to the protocol.
* Patients who have a diagnosis or history suggestive of chemical dependence, or drug-induced toxic psychosis in the preceding 6 months; diagnosis or history of abuse (except for nicotine and caffeine) within the past 3 months, or a clinical presentation possibly confounded by the use of recreational drugs or alcohol.
* Patients who have a positive urine drug screen (at the screening visit). If opiates are positive at screening and clearly due to the use of pain killing medication, the patient may be re screened after the medication has been discontinued and enrolled in the study if urine drug screen is negative.
* Note: Occasional users of recreational drugs other than cocaine, amphetamines, hallucinogens, or parenteral drugs may be recruited. Patients who are dependent on nicotine, caffeine, or theophylline are allowed to enter the study.
* Patients who are mentally disabled (moderate to severe).
* Patients who have had a history of being in a coma for more than 24 hrs.
* Patients who have had thoughts of committing suicide within 6 months prior to screening or at baseline or suicide behaviors within 2 years prior to screening or at baseline.
* Patients thought to be of imminent risk of harm to others or in imminent legal difficulty.
* Patients under any form of legal compulsion to remain hospitalized or undergo treatment or assessment.
* Patients who have any disability that prevent them from completing any of the study requirements.
* Patients with a known clinically significant ECG abnormality including PR interval >240 msec, QRS complex >110 msec, QTcF >=450 msec, or congenital long QT syndrome based on central ECG reading results
* Treatment naive, first episode patients,
* Patients taking iloperidone at the screening visit or with a known hypersensitivity to drugs chemically related to benzioxazoles.
* Note: Active medical conditions that are minor or well-controlled are not exclusionary if they do not affect risk to the patient or the study results.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 635 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (25):
  - Vanda Investigative Site, Anaheim, California
  - Vanda Investigative Site, Bellflower, California
  - Vanda Investigative Site, Costa Mesa, California
  - Vanda Investigative Site, Escondido, California
  - Vanda Investigative Site, La Habra, California
  - Vanda Investigative Site, Oceanside, California
  - Vanda Investigative Site, Orange, California
  - Vanda Investigative Site, Pico Rivera, California
  - Vanda Investigative Site, Riverside, California
  - Vanda Investigative Site, San Diego, California
  - Vanda Investigative Site, Santa Ana, California
  - Vanda Investigative Site, Melbourne, Florida
  - Vanda Investigative Site, Miami, Florida
  - Vanda Investigative Site, Oakland Park, Florida
  - Vanda Investigative Site, Atlanta, Georgia
  - Vanda Investigative Site, St Louis, Missouri
  - Vanda Investigative Site, Nashua, New Hampshire
  - Vanda Investigative Site, Marlton, New Jersey
  - Vanda Investigative Site, Brooklyn, New York
  - Vanda Investigative Site, Staten Island, New York
  - Vanda Investigative Site, Hickory, North Carolina
  - Vanda Investigative Site, Beachwood, Ohio
  - Vanda Investigative Site, Philadelphia, Pennsylvania
  - Vanda Investigative Site, Irving, Texas
  - Vanda Investigative Site, Salt Lake City, Utah
- India (11):
  - Vanda Investigative Site, Ahmedabad, Gujarat
  - Vanda Investigative Site, Madhava Nagar, Karnataka
  - Vanda Investigative Site, Mangalore, Karnataka
  - Vanda Investigative Site, Mysore, Karnataka
  - Vanda Investigative Site, Nashik, Maharashtra
  - Vanda Investigative Site, Pune, Maharashtra
  - Vanda Investigative Site, Jaipur, Rajasthan
  - Vanda Investigative Site, Madurai, Tamil Nadu
  - Vanda Investigative Site, Kanpur, Uttar Pradesh
  - Vanda Investigative Site, Lucknow, Uttar Pradesh
  - Vanda Investigative Site, Varanasi, Uttar Pradesh
- Ukraine (17):
  - Vanda Investigative Site, Kerch, AR Crimea
  - Vanda Investigative Site, Yevpatoria, AR Crimea
  - Vanda Investigative Site, Chernihiv
  - Vanda Investigative Site, Dnipropetrovsk
  - Vanda Investigative Site, Donetsk
  - Vanda Investigative Site, Ivano-Frankivsk
  - Vanda Investigative Site, Kharkiv
  - Vanda Investigive Site, Kharkiv
  - Vanda Investigative Site, Kyiv
  - Vanda Investigative Site, Luhansk
  - Vanda Investigative Site, Odesa
  - Vanda Investigative Site, Poltava
  - Vanda Investigative Site, Simferopol
  - Vanda Investigative Site, Stepanovka
  - Vanda Investigative Site, Ternopil
  - Vanda Investigative Site, Uzhhorod
  - Vanda Investigative Site, Vinnytsia

REFERENCES:
- [Result] Weiden PJ, Manning R, Wolfgang CD, Ryan JM, Mancione L, Han G, Ahmed S, Mayo MG. A Randomized Trial of Iloperidone for Prevention of Relapse in Schizophrenia: The REPRIEVE Study. CNS Drugs. 2016 Aug;30(8):735-47. doi: 10.1007/s40263-016-0345-4. PMID 27379654

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 635 patients were enrolled and received iloperidone in the Cross-Titration Phase and entered Stabilization Phase. A total of 303 were randomized and received either iloperidone (n=153) or placebo (n=150) in the Double-Blind Relapse Prevention Phase.
Groups:
- Iloperidone: After meeting all entry criteria, completing a 1-week open-label iloperidone titration period (up to 12 mg/day), followed by a 14-24 week open-label iloperidone flexible dose-stabilization period (up to 24 mg/day), patients in this arm were randomized to iloperidone (flexible dosing 8-24 mg/day). Post-randomization double-blind study medication was administered orally twice daily for up to 26 weeks to evaluate relapse prevention. Subsequently, during the extension period, after a 1-week mock double-blind titration, open-label iloperidone (8-24 mg/day) was administered for up to 51 weeks to evaluate long-term safety.
- Placebo: After meeting all entry criteria, completing a 1-week open-label iloperidone titration period (up to 12 mg/day), followed by a 14-24 week open-label iloperidone flexible dose-stabilization period (up to 24 mg/day), patients in this arm were randomized to matching placebo. Post-randomization double-blind study medication was administered orally twice daily for up to 26 weeks to evaluate relapse prevention.
Period: Cross-Titration and Stabilization Phase
Arm/Group | Iloperidone | Placebo
Started | 635 | 0
Completed | 309 | 0
Not Completed | 326 | 0
Not completed — Withdrawal by Subject | 107 | 0
Not completed — Adverse Event | 92 | 0
Not completed — Administrative problems | 30 | 0
Not completed — Lack of Efficacy | 28 | 0
Not completed — Abnormal Laboratory Value | 25 | 0
Not completed — Lost to Follow-up | 24 | 0
Not completed — Protocol Violation | 13 | 0
Not completed — Abnormal test | 6 | 0
Not completed — Death | 1 | 0
Period: Double-blind Relapse Prevention Phase
Arm/Group | Iloperidone | Placebo
Started | 153 | 150
Completed | 76 | 102
Not Completed | 77 | 48
Not completed — Administrative problems | 45 | 29
Not completed — Withdrawal by Subject | 14 | 10
Not completed — Lost to Follow-up | 6 | 4
Not completed — Adverse Event | 5 | 0
Not completed — Abnormal Laboratory Value | 4 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Abnormal test | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Iloperidone: oral, open-label titration up to 12 mg for 1-week followed by open-label flexible dosing (8-24 mg/day), followed by double-blind 8-24 mg/day dosing for 26 weeks
- Placebo: oral, matching placebo administered during double-blind phase for up to 26 weeks
- Total: Total of all reporting groups
Arm/Group | Iloperidone | Placebo | Total
Number analyzed (Participants) | 153 | 150 | 303
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (11.3) | 38.2 (11.1) | 38.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 68 | 125
  Male | 96 | 82 | 178
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 74 | 77 | 151
  Black | 31 | 28 | 59
  Asian | 38 | 40 | 78
  Pacific Islander | 1 | 0 | 1
  Other | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse or Impending Relapse
Description: Relapse or impending relapse was defined as any of the following: hospitalization due to worsening of schizophrenia; increase (worsening) of the PANSS total score of greater than or equal to 30% from randomization, PANSS total score confirmed at a second visit conducted within 1-7 days; clinically significant emergent or worsening suicidal, homicidal, or aggressive behavior; a CGI-Improvement (CGI-I) score of 6 (much worse) or 7 (very much worse) after randomization; a dose increase in study medication or a need for additional open-label antipsychotic treatment.
Time Frame: Up to 26 weeks post-randomization
Population: Two subjects lost to follow-up after randomization were excluded from the analysis population.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Iloperidone: oral, flexible dosing 8-24 mg/day given bid
- Placebo: oral, matching placebo given bid
Arm/Group | Iloperidone | Placebo
Number analyzed (Participants) | 151 | 150
Days | NA [NA to NA] — The median relapse free time could not be estimated as the Kaplan-Meier probability estimate of relapse over the 26-week double-blind period did not exceed 50% (i.e. the median, lower and upper limit of 95% CI was not estimable due to low number of participants with events). | 99 [57 to 122]
Statistical Analysis 1: Comparison: Iloperidone vs Placebo; Test type: Superiority; p < 0.0001, Log Rank; Cox Proportional Hazard = 5.2, 95% CI 2-sided [3.2 to 8.4]

2. Secondary Outcome: PANSS Total Score, Change From Baseline to Last Visit
Description: The 30-item Positive and Negative Syndrome Scale (PANSS) was developed to assess the severity of symptoms of schizophrenia. The PANSS items are divided into positive, negative, and general psychopathology factors. All items were rated on a scale of 1 (absent) to 7 (extremely severe). The PANSS total score (or rating) is the sum of all 30 PANSS items taken together (the sum of its 3 subscales), with a maximum score of 210. Change from baseline is calculated as post value minus baseline value. A negative change indicates improvement.
Time Frame: Up to 26 weeks post-randomization
Population: Data presented are FAS (Full Analysis set) LOCF (last observation carried forward) Change From DBRP (Double-Blind Relapse Prevention) Baseline to RP Completion. RP Completion visit includes observations from last visit during DBRP period for patients who completed the study or RP Completion visit for patients who discontinued the DBRP phase and not included in previous scheduled visit.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Iloperidone | Placebo
Number analyzed (Participants) | 150 | 149
units on a scale | 1.1 (1.12) | 12.4 (1.15)
Statistical Analysis 1: Comparison: Iloperidone vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — P-value is based on an ANCOVA model with treatment and site as main effects and DBRP baseline as a covariate

3. Secondary Outcome: CGI-S, Last Visit
Description: The 7-item Clinical Global Impression of Severity (CGI-S) scale was developed to assess the overall, absolute degree of illness at any point in time. A rating of 1 is equivalent to "normal, not at all ill," and a rating of 7 is equivalent to "among the most extremely ill patients."
Time Frame: Up to 26 weeks post-randomization
Population: Data presented are FAS (Full Analysis set) OC (observed cases), as this measure does not include a baseline assessment; RP Completion visit includes observations from last visit during DBRP period for patients who completed the study and RP Completion visit that could not be remapped to a previous scheduled visit for patients who discontinued the DBRP phase.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Iloperidone | Placebo
Number analyzed (Participants) | 112 | 105
units on a scale | 3.0 (0.89) | 3.6 (1.11)

4. Secondary Outcome: SDS Total Score, Change From Baseline to Last Visit
Description: The Sheehan Disability Scale (SDS) a self-reported measure that was developed to assess functional impairment in 3 inter-related domains (i.e., work/school, social, and family life). It is a 10-point visual analog scale with 0 being not impaired at all and 10 extremely impaired. Change from baseline is calculated as post value minus baseline value. A negative change indicates improvement.
Time Frame: Up to 26 weeks post-randomization
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Iloperidone | Placebo
Number analyzed (Participants) | 142 | 128
units on a scale | -0.2 (0.54) | 1.8 (0.61)
Statistical Analysis 1: Comparison: Iloperidone vs Placebo; Test type: Superiority; p = 0.0062, ANCOVA — P-value is based on an ANCOVA model with treatment and site as main effects and DBRP baseline as a covariate

ADVERSE EVENTS:
Time Frame: Cross-Titration Phase (1 week) and Stabilization Phase (14-24 weeks); Relapse-prevention phase (up to 26 weeks)
Description: For each phase, i.e. Cross-titration/Stabilization Phase and Relapse-prevention Phase, the safety population included all enrolled or randomized patients who received at least 1 dose of study drug during the corresponding phase. For the Relapse-prevention Phase, in case of a treatment error, patients were analyzed according to the treatment received.
Groups:
- Iloperidone (Cross-titration and Stabilization Phase): During the 1 week Cross-titration phase, patients were titrated up to 12 mg/d open-label iloperidone orally twice a day. The prior antipsychotic was discontinued by day 4. During the 14 to 24 week Stabilization Phase, the dose could be modified within a permitted range of a total daily dose of 8-24 mg/d.
- Iloperidone (Relapse-prevention Phase): Patients received 8 to 24 mg/d iloperidone orally twice a day for up to 26 weeks.
- Placebo (Relapse-prevention Phase): Patients received placebo orally twice a day for up to 26 weeks.
Arm/Group | Iloperidone (Cross-titration and Stabilization Phase) | Iloperidone (Relapse-prevention Phase) | Placebo (Relapse-prevention Phase)
All-Cause Mortality (participants affected / at risk) | 1/629 | 1/151 | 0/150
Serious Adverse Events (participants affected / at risk) | 21/629 | 6/151 | 4/150
Other Adverse Events (participants affected / at risk) | 244/629 | 16/151 | 30/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iloperidone (Cross-titration and Stabilization Phase) (N=629) | Iloperidone (Relapse-prevention Phase) (N=151) | Placebo (Relapse-prevention Phase) (N=150)
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Arthritis viral (Infections and infestations) | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 9 | 2 | 2
Acute psychosis (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 0
Alcoholism (Psychiatric disorders) | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Priapism (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Iloperidone (Cross-titration and Stabilization Phase) (N=629) | Iloperidone (Relapse-prevention Phase) (N=151) | Placebo (Relapse-prevention Phase) (N=150)
Schizophrenia (Psychiatric disorders) | 8 | 1 | 13
Insomnia (Psychiatric disorders) | 35 | 3 | 7
Dizziness (Nervous system disorders) | 73 | 4 | 4
Headache (Nervous system disorders) | 40 | 3 | 5
Weight Increased (Investigations) | 34 | 2 | 4
Nausea (Gastrointestinal disorders) | 32 | 2 | 0
Somnolence (Nervous system disorders) | 52 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 43 | 0 | 0

LIMITATIONS AND CAVEATS:
The primary limitation of the study design is that the length of the placebo-controlled phase of the study lasted for only 6 months. However, ethical considerations around the use of placebo in this patient population necessarily informed the study design. While the flexible-dosing regimen in this study allowed for a more real-world experience, it also prevented the assessment of dose-response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pooled site data analysis is restricted to publication by consent of steering committee. PI is restricted from presenting or publishing independently on their own site data until the expiration of eighteen (18) months from the completion of the Clinical Trial or as otherwise noted in the Investigator's clinical trial agreement.